CLINICAL TRIAL: NCT05592015
Title: A Phase II Study Evaluating the Efficacy of Ruxolitinib in Patients With T-Cell Large Granular Lymphocytic Leukemia (T-LGLL)
Brief Title: Ruxolitinib for the Treatment of T-Cell Large Granular Lymphocytic Leukemia
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Jonathan Brammer (Other)
Responsible Party: Sponsor-Investigator, Jonathan Brammer, Principal Investigator, Ohio State University Comprehensive Cancer Center
Organization: Ohio State University Comprehensive Cancer Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OSU-21336; NCI-2022-02385 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2022-04-18; First posted 2022-10-24 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: T-Cell Large Granular Lymphocyte Leukemia
MeSH Terms: conditions — Leukemia, Large Granular Lymphocytic | interventions — ruxolitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (ruxolitinib) (Experimental): Patients receive ruxolitinib PO BID on days 1-28. Cycles repeat every 28 days for 12 months in the absence of disease progression or unacceptable toxicity. Patients who achieve a response (CR or PR) may receive an additional 12 months of ruxolitinib, for a maximum of 24 months.
  Interventions: Drug: Ruxolitinib

INTERVENTIONS:
Drug: Ruxolitinib — Given PO
  Other Names: INCB-18424; INCB18424; Jakafi; Oral JAK Inhibitor INCB18424

SUMMARY:
This phase II trial tests whether ruxolitinib works to shrink tumors in patients with T-cell large granular lymphocyte leukemia. Ruxolitinib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Determine the overall response rate (ORR) of ruxolitinib in patients with T-cell large granular lymphocytic leukemia (T-LGLL) as compared to historical controls.

SECONDARY OBJECTIVES:

I. Rate of conversion from PR at 4 months to CR at 8 and 12 months (at full ruxolitinib dosage).

II. Rate of molecular remission (T-cell receptor [TCR] clearance, STAT3 mutation clearance) at 4, 8, 12 months.

III. Incidence of grade III/IV toxicities (at full ruxolitinib dosage). IV. Quality of life using the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30 (EORTC QLQ-C30), Health Assessment Questionnaire Disability Index (HAQDi), and Short Form (SF)-36 questionnaire at baseline, 5 months, and every 6 months during response follow up for up to 12 months.

EXPLORATORY OBJECTIVE:

I. Objective benefit (OB) rate at 4 months defined as a patient that had improvement in their cytopenias, transfusion dependence but not attaining a partial response (PR).

II. Leukemia-free survival III. Progression-free survival

OUTLINE:

Patients receive ruxolitinib orally (PO) twice daily (BID) on days 1-28. Cycles repeat every 28 days for 12 months in the absence of disease progression or unacceptable toxicity. Patients who achieve a response (CR or PR) may receive an additional 12 months of ruxolitinib, for a maximum of 24 months. Additionally, patients undergo blood sample collection throughout study.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older and able to swallow pills
* Diagnosis of T-LGLL defined as: LGL cell population meeting diagnostic criteria (defined as CD3+CD8+ cell population >650/mm3 or CD3+CD8+CD57+ population >500/mm3 or LGL cell population with other immunophenotype that includes co-expression of CD3+, CD8+, CD57+ with >500 cells/mm3 and the presence of a clonal T-cell receptor (within 1 month of diagnosis or relapse). This also includes patients with rare T-LGLL variants include CD4+ T-LGLL, and gamma/delta T-LGLL which can be CD4- and CD8-), though patients still must have the presence of a clonal T-cell receptor within 1 month of diagnosis or relapse. Note: patients with MDS-like T-LGLL may be included with PI approval even if CD3+CD8+ cell population is < 650/mm^3, though +TCR is required. Natural-Killer (NK) LGL is also permitted, provided there is a clonal NK-cell population noted with > 500 cells/mm^3
* Untreated T-LGLL or failed at least one line of frontline therapy;
* Patients must be off treatment for at least 14 days or 5 half-lives, whichever is longer
* Require Treatment for T-LGLL (one or more required)

  * Symptomatic anemia with hemoglobin < 10 g/dL
  * Transfusion-dependent anemia
  * Neutropenia with absolute neutrophil count (ANC) < 500/mm^3
  * Neutropenia with ANC < 1500/mm^3 with recurrent infections
* Platelet count > 50 x 10^9/L. Platelet transfusion may be utilized to meet inclusion criteria, as long as the platelet count remains >50,000/uL within 5 days of last transfusion. Note: Patients with platelets <100 x 109/L and renal impairment are not permitted to enroll to the study. Renal impairment is defined as creatinine clearance (CrCl) < 90 mL/min.
* Serum creatinine =< 2 x the upper limit of normal (ULN)
* - Estimated glomerular filtration rate (eGFR) => 30 mL/min using the Modification of Diet in Renal Disease (MDRD) equation (multiplying eGFR by each subjects Body Surface Area [BSA])
* Total bilirubin =< 1.5 x ULN (patients with Gilbert's syndrome with a bilirubin > 1.5 x ULN permitted)
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) =< 2.5 x ULN
* Alkaline phosphatase (ALP) =< 2.5 x ULN
* Eastern cooperative oncology group (ECOG) performance status =< 2
* Men and women of reproductive potential must agree to follow accepted birth control methods for the duration of the study. Female subject is either post-menopausal or surgically sterilized or willing to use an acceptable method of birth control (i.e., a hormonal contraceptive, intra-uterine device, diaphragm with spermicide, condom with spermicide, or abstinence) for the duration of the study treatment until 5 half-lives have passed. Male subject agrees to use an acceptable method for contraception for the duration of the study treatment until 5 half-lives have passed.
* Able to sign informed consent

Exclusion Criteria:

* Absolute neutrophil count (ANC) less than 100/mm^3. Note: granulocyte colony-stimulating factor (G-CSF) may be utilized to enable patients to meet inclusion criteria, as long as the ANC remains above 100/mm^3 for 5 days after administration of last growth-factor.
* Active infection requiring ongoing anti-microbial treatment. Patients with human immunodeficiency virus (HIV), positive hepatitis B surface antigen or hepatitis C antibody will be excluded. Patients with tuberculosis risk factors will be required to undergo quantiferon testing and/or purified protein derivative (PPD) testing with a negative result prior to entering the study.
* Concurrent immune-suppressive therapy (prednisone or equivalent up to 20 mg permitted to treat LGLL symptoms, but must be weaned within one month of initiation of trial drug). Patients on stable, chronic prednisone =< 10 mg for rheumatologic/autoimmune conditions are exempted from this requirement. They may enroll on the study
* Active, concurrent malignancy unless deemed related to T-LGLL by principal investigator (PI). Early stage skin cancers, prostate cancer, permitted if under no active therapy
* For females of childbearing potential: Positive pregnancy test or lactating
* Unstable angina or myocardial infarction within the past 2 months
* Chronic obstructive pulmonary disease or other interstitial lung disease in active exacerbation
* Cirrhosis
* For any strong CYP3A4 inhibitors deemed a moderate or severe risk of interaction with ruxolitinib, a wash-out period of 14 days, or 5 half-lives, whichever is longer, is needed prior to starting ruxolitinib
* Given the CYP3A4 inhibition potential of grapefruit, grapefruit juice, Seville orange juice, pomelos, and starfruits, patients will need to refrain from these foods/drinks for 14 days prior to initiation of therapy, and throughout the study period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-05-03 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (ORR) | Up to 12 months
  The ORR will be calculated as the proportion of patients who achieve a response to therapy divided by the total number of evaluable patients. An evaluable patient is defined as an eligible patient who has received at least four months of therapy with ruxolitinib. All evaluable patients will be included in calculating the ORR for the study along with corresponding 95% binomial confidence intervals (CIs) (assuming that the number of patients who respond is binomially distributed). Additional outcomes including rates of conversion from PR at 4 months to CR at 8 and 12 months on full dose ruxolitinib, and rate of molecular remission (TCR clearance, STAT3 mutation clearance) at 4, 8, 12 months on full dose ruxolitinib will also be reported as proportions with 95% binomial CIs.

SECONDARY OUTCOMES:
Incidence of treatment-emergent adverse events | Up to 12 months
  Treatment-emergent adverse events will be reported overall and by toxicity grade.
Leukemia-free survival (LFS) | From first response until disease progression, death, or censoring (if alive and disease-free at the end of follow-up), assessed up to 12 months
  Kaplan Meier curves will be generated and the median LFS and 95% CIs will be reported.
Patient quality-of-life (QOL) EORTC | Up to 12 months
  Will be assessed via responses to the European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire at baseline, 5 months, and 1 year on study. Changes in QOL will be calculated from the differences in scores between baseline and 5 months, baseline and 1 year, and 5 months and 1 year, for each patient. The proportions of patients who had improvement in QOL scores between time points will be compared between responding patients and non-responding patients, patients with and without rheumatologic disease, and between patients classified as having an objective benefit and patients who did not have an objective benefit. Mean changes in patient QOL between time points will also be reported.
Patient quality-of-life (QOL) QLQ-C30 | Up to 12 months
  Will be assessed via responses to the European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire-Core 30 given at baseline, 5 months, and 1 year on study. Changes in QOL will be calculated from the differences in scores between baseline and 5 months, baseline and 1 year, and 5 months and 1 year, for each patient. The proportions of patients who had improvement in QOL scores between time points will be compared between responding patients and non-responding patients, patients with and without rheumatologic disease, and between patients classified as having an objective benefit and patients who did not have an objective benefit. Mean changes in patient QOL between time points will also be reported.
Patient quality-of-life (QOL) HAQDi | Up to 12 months
  Will be assessed via responses to the European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire-Health Assessment Questionnaire-Disability Index questionnaires given at baseline, 5 months, and 1 year on study. Changes in QOL will be calculated from the differences in scores between baseline and 5 months, baseline and 1 year, and 5 months and 1 year, for each patient. The proportions of patients who had improvement in QOL scores between time points will be compared between responding patients and non-responding patients, patients with and without rheumatologic disease, and between patients classified as having an objective benefit and patients who did not have an objective benefit. Mean changes in patient QOL between time points will also be reported.
Patient quality-of-life (QOL) SF-36 | Up to 12 months
  Will be assessed via responses to the European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire-Short Form-36 given at baseline, 5 months, and 1 year on study. Changes in QOL will be calculated from the differences in scores between baseline and 5 months, baseline and 1 year, and 5 months and 1 year, for each patient. The proportions of patients who had improvement in QOL scores between time points will be compared between responding patients and non-responding patients, patients with and without rheumatologic disease, and between patients classified as having an objective benefit and patients who did not have an objective benefit. Mean changes in patient QOL between time points will also be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Brammer, MD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (3):
- United States (3):
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu